CLINICAL TRIAL: NCT01324726
Title: Sites of Colonization in Hospitalized Patients With Infections Caused by Extended-Spectrum Beta-Lactamase Producing Escherichia Coli and Klebsiella Pneumoniae
Brief Title: Colonization With Extended-Spectrum Beta-Lactamase (ESBL)-Producing Organisms
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Zeina Kanafani, Doctor, Internal Medicine, American University of Beirut Medical Center
Other Study IDs: IM.ZK.05
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Escherichia Coli Infections; Klebsiella Pneumonia
Keywords: Bacterial colonization; Extended spectrum beta lactamase producing organisms
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cultures of urine, nasopharynx, rectum, skin, and wounds
Oversight: Data Monitoring Committee: No

SUMMARY:
There has been a great increase in the incidence of infections caused by bacteria that are resistant to antibiotic agents. Many of these infections result in worse outcomes of patients and increased costs to the healthcare system. The study aims to survey two germs that are resistant to a wide range of antibiotics used today. The investigators are particularly interested in studying the potential to stop the spread and prevent outbreaks of these germs through contact isolation of patients affected by these germs. Patients will be included in the study if they have an antibiotic resistant infection caused by any of the 2 bacteria: E. coli and K. pneumoniae. The research team will then perform rectal, skin (armpit, groin, umbilicus), throat, urine, and, if applicable, wound cultures to determine other sites where the germ may be present but not causing an infection. The study coordinator will furthermore examine the patient's medical record and conduct a short interview in order to evaluate specific information about the bacteria that have been recovered. This research does not involve any interventions beyond collection of specimens and there are no added risks to the patients from the conduction of the study. Neither will there be a benefit at the patient level. The benefit will be at the level of the patient population, i.e. at a larger scale once the information collected is analyzed. Only the principal investigator and study coordinators will have access to all patient-specific information. Once all information is collected, all patient identifiers, such as name and medical record number, will be deleted.

DETAILED DESCRIPTION:
The rising incidence of infections caused by extended-spectrum beta-lactamase (ESBL) producing Enterobacteriaceae is of worldwide dimensions, particularly in developing countries. At the American University of Beirut Medical Center (AUB-MC), the proportion of ESBL producing E. coli (ESBL-EC) and K. pneumoniae (ESBL-KP) strains has risen from 2.5% and 9.8% to 22% and 27%, respectively between 1999 and 2008. The rapid spread of these multi drug resistant pathogens prompted the study of factors aiming at limiting the ongoing transmission of these organisms. Infection control interventions, such as contact isolation of infected patients, have been used to control outbreaks of infections caused by ESBL producing organisms in settings where the pathogens were isolated from rectal and axillary samples, as well as from upper respiratory tract secretions. These few reports raise concern for colonization of infected patients at sites other than the primary site of infection. Colonization in the absence of outbreaks has so far not been looked at systematically, especially in a high-endemicity area such as Lebanon. The present study ultimately aims at assessing the usefulness of placing patients with ESBL-EC and ESBL-KP infections on contact isolation during their hospital stay, and whether this practice would limit the spread of such infections. This is a prospective study screening hospitalized patients with ESBL-EC and ESBL-KP infections for colonization with the same organism at sites other than the primary site of infection through cultures of the rectum, skin, nasopharynx, urine and, if applicable, wounds. Cases will be identified through the Clinical Microbiology Laboratory at AUBMC and study subjects will be enrolled according to the inclusion/exclusion criteria. In addition to cultures of multiple body sites, molecular analysis will be performed on the isolated ESBL-producing strains to identify clonal relatedness. Cultures will be repeated monthly for a period of 6 months. The sample size is estimated at 100 patients over a two year period. The results of this study will have implications on infection control practices and will constitute a prerequisite for further studies in the future.

The objective of this proposal is to evaluate the extent of colonization with ESBL-EC and ESBL-KP in hospitalized patients with active infections and designing recommendations accordingly.

The specific aims include:

1. Identify hospitalized patients with infections due to ESBL-producing organisms at a primary site
2. Screen patients for colonization with ESBL-producing organisms at body sites other than the primary site of infection through cultures of:

   * Rectum
   * Skin (axillae, groin, umbilicus)
   * Nasopharynx
   * Urine
   * Wound (if applicable)
3. Perform susceptibility testing on all the collected isolates to detect ESBL-EC and ESBL-KP
4. Perform molecular testing on ESBL-producing pathogens isolated from sites of colonization and compare them to the organisms recovered from the primary site in order to identify clonal relatedness
5. Perform follow up cultures from the above mentioned sites after treatment for the primary infection is completed to determine duration of colonization
6. Draw conclusions regarding extent of colonization with ESBL-producing organisms in hospitalized patients with a primary infection and to evaluate infection control implications (particularly with respect to placing patients on isolation precautions)

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients with infection caused by ESBL-EC or ESBL-KP
2. Type of infections:

   * Urinary tract infections
   * Respiratory tract infections
   * Skin and skin structure infections
   * Bloodstream infections

Exclusion Criteria:

1. Age < 18 years
2. Infection with the same antibiotic-resistant organism within the preceding year
3. Intake of effective antibiotics based on susceptibility testing for longer than 48 hours at the time of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cultures from clinical specimens growing ESBL-EC and ESBL-KP will be identified through the Clinical Microbiology Laboratory at AUBMC. Patients will be selected for enrollment according to the inclusion and exclusion criteria previously set. Permission from the patient's primary physician will be sought at the time of identification before approaching the patient.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of colonization sites | 3 days
  This describes the number of body sites at which the patient is colonized other than the primary site of infection.

SECONDARY OUTCOMES:
Time until clearance of colonization | 6 months
  This describes the time until various body sites become clear of colonizing pathogens.

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Beyrouth, Lebanon